CLINICAL TRIAL: NCT06631703
Title: Effect of Oropharyngeal Colostrum Administration on Early Feeding Skills in Premature Infants
Brief Title: Oropharyngeal Colostrum Administration in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sinem Yalnızoglu Caka, Assoc. Prof., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20222503; Kocaeli University (Other: Kocaeli University)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Oral Colostrum Administration; Early Feeding Skills; Transition to Oral Feeding
Keywords: Premature infant; oral colostrum; feeding skills
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: This single-blind, randomized, controlled study was conducted with a pre-test and post-test control group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group receiving Oral Colostrum Administiration (Experimental): In the premature infants in the intervention group in which oropharyngeal colostrum was administered, the application was performed as follows: The oropharyngeal colostrum administration technique consists of slowly inserting a sterile 1 mL syringe without a needle with the tip of the syringe into the baby's mouth along the right buccal mucosa (0.1 mL) towards the oropharynx, then moving the syringe towards the inside of the cheeks and on the tongue, and repeating the same procedure on the left buccal mucosa (0.1 mL) without removing it (slow administration in approximately 1 minute). The routine feeding procedure was then continued.
  Interventions: Other: Group receiving Oral Colostrum Administiration
- Routine Feeding Care (No Intervention): According to the NICU guidelines, The control group continued to receive the routine feeding plan. Within the scope of the study, infants in both groups received colostrum, the only difference being the route of administration. The control group received colostrum by gavage, and the study group received colostrum using an oropharyngeal route.

INTERVENTIONS:
Other: Group receiving Oral Colostrum Administiration — Description: Colostrum secreted in the first 3-5 days was oropharyngeal administered to the intervention group by withdrawing 0.2 ml of colostrum to be taken from the mother with the help of an insulin injector every three hours before each feeding meal in accordance with the literature.In the premature infants in the intervention group in which oropharyngeal colostrum was administered, the application was performed as follows: The oropharyngeal colostrum administration technique consists of slowly inserting a sterile 1 mL syringe without a needle with the tip of the syringe into the baby's mouth along the right buccal mucosa (0.1 mL) towards the oropharynx, then moving the syringe towards the inside of the cheeks and on the tongue, and repeating the same procedure on the left buccal mucosa (0.1 mL) without removing it (slow administration in approximately 1 minute). The routine feeding procedure was then continued
  Arms: Group receiving Oral Colostrum Administiration

SUMMARY:
this study aimed to determine the effect of oropharyngeal colostrum administration on premature newborns on early feeding cues and transition time to full oral feeding.

DETAILED DESCRIPTION:
Breastfeeding has immunologic, nutritional, and neurodevelopmental benefits for premature infants. Follow-up of premature infants in the Neonatal Intensive Care Unit (NICU) for observation and treatment due to immature gestational age, organ or system diseases, and inadequate oral sucking power cause physical and psychological separation of mother and infant, and this is an essential factor leading to breastfeeding failure. Despite the abundant evidence in the literature for the benefits of breast milk and especially colostrum for premature infants, breastfeeding and lactation rates are still very low in this vulnerable population due to poor sucking/swallowing/respiratory coordination.

Although the development of oral feeding skills in premature infants is a challenge for health professionals and parents, oral feeding skills are one of the critical indicators for the discharge of premature infants. Although motor activities such as sucking, swallowing, and breathing are known to be present in the prenatal period, it is not known precisely when this coordination is achieved at the earliest after birth. Approximately 40% of premature infants have difficulty transitioning from enteral to oral feeding. A systematic review showed that premature infants experience problems with oral feeding in the first four years of life, with a prevalence of 42%. Physiological intervention methods that support the transition of premature infants to oral feeding include non-nutritive sucking, oral-motor stimulation, and oral care with colostrum or breast milk. Oropharyngeal colostrum administration is an intervention method reported to activate the digestive hormones of minimal enteral feeding, encourage feeding, accelerate the maturation of the gastrointestinal system, and shorten the transition to full oral feeding with positive stimulation. When the literature is examined, it is reported that premature infants fed with colostrum from the NICU also have increased breastfeeding continuity after discharge. The most crucial difference between our study and the studies available in the literature is related to how oropharyngeal administered colostrum affects the infant's early feeding cues (coordination of sucking-swallowing and respiration during feeding) and how much it accelerates/shortens the transition to oral feeding. In the literature, no study is similar to our study examining how oropharyngeal colostrum administration affects this process in the transition to full oral feeding using a measurement tool on the subject.

ELIGIBILITY:
Inclusion Criteria:

* The gestational week at the time of delivery is between 260-33+6 gestational weeks, determined according to the mother's last menstrual date and obstetric evaluation results.
* Started feeding with an orogastric catheter, in the process of transition from catheter feeding to oral feeding
* Meeting early feeding readiness criteria (stable respiration and oxygen saturation during feeding, responsiveness to perioral/oral stimulation and licking, etc.)
* 750 g or more during the study
* Stable vital signs (respiratory rate <60/min, heart rate 140-185 beats/min, axillary temperature 36.5-37.4°C) (Acunaş et al., 2018)
* NICU admission ≤ 24 hours of life; protocol can be started within 72 hours,
* No muscle relaxants, sedatives, or severe neurological disease
* Allowing parents of premature infants

Exclusion Criteria:

* Congenital or chromosomal anomalies, lack of cardiorespiratory stabilization, birth asphyxia (cord ph/arterial ph <7. 0), twin or more multiple births, intrauterine growth retardation, necrotizing enterocolitis, pneumothorax, skull fracture, severe atelectasis, circulatory disorder, severe sepsis, having a chest tube, having a history of pathologic jaundice, having a history of antenatal gastrointestinal system disease, born with cleft palate/lip, born to mothers with confirmed chorioamnionitis were excluded.

Ages: 26 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Early Feeding Skills Assessment | 10 days
  Evaluation will begin with oral colostrum administration to premature infants. The tool allows the assessment of preterm infants' readiness for oral feeding and oral feeding skills, the observation of symptoms associated with problem feeding, and the planning of feeding interventions targeting areas where the infant has difficulty or needs support during the transition to oral feeding. Both the revised EFS and the Turkish version of the EFS include 19 items in 5 subscales. These subscales are respiratory regulation, oral-motor function, swallowing coordination, feeding participation, and physiological stability.

SECONDARY OUTCOMES:
Full oral feeding time | 20 days
  The days of transition to full oral feeding of the babies in the experimental and control groups will be evaluated throughout the application.
Weight gain | 10 days
  The weight gain processes of the babies in the experimental and control groups will be evaluated throughout the application with the scales used in the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Sümeyra Topal, Kahramanmaraş, Dulkadiroğlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nasuf AWA, Ojha S, Dorling J. Oropharyngeal colostrum in preventing mortality and morbidity in preterm infants. Cochrane Database Syst Rev. 2018 Sep 7;9(9):CD011921. doi: 10.1002/14651858.CD011921.pub2. PMID 30191961
- [Background] Manerkar S, Kalamdani P, Patra S, Kalathingal T, Mondkar J. Improving Early Colostrum Feeding in a Tertiary Neonatal Intensive Care Unit: A Quality Improvement Initiative. Breastfeed Med. 2022 Feb;17(2):143-148. doi: 10.1089/bfm.2021.0173. Epub 2021 Nov 2. PMID 34726511
- [Background] Li L, Liu L, Chen F, Huang L. Clinical effects of oral motor intervention combined with non-nutritive sucking on oral feeding in preterm infants with dysphagia. J Pediatr (Rio J). 2022 Nov-Dec;98(6):635-640. doi: 10.1016/j.jped.2022.02.005. Epub 2022 May 13. PMID 35569569
- [Background] Kumar J, Meena J, Ranjan A, Kumar P. Oropharyngeal application of colostrum or mother's own milk in preterm infants: a systematic review and meta-analysis. Nutr Rev. 2023 Sep 11;81(10):1254-1266. doi: 10.1093/nutrit/nuad002. PMID 36718589
- [Background] Grundt H, Tandberg BS, Flacking R, Drageset J, Moen A. Associations Between Single-Family Room Care and Breastfeeding Rates in Preterm Infants. J Hum Lact. 2021 Aug;37(3):593-602. doi: 10.1177/0890334420962709. Epub 2020 Oct 9. PMID 33035125
- [Background] Glass KM, Greecher CP, Doheny KK. Oropharyngeal Administration of Colostrum Increases Salivary Secretory IgA Levels in Very Low-Birth-Weight Infants. Am J Perinatol. 2017 Dec;34(14):1389-1395. doi: 10.1055/s-0037-1603655. Epub 2017 Jun 2. PMID 28575910
- [Background] Zhang Y, Ji F, Hu X, Cao Y, Latour JM. Oropharyngeal Colostrum Administration in Very Low Birth Weight Infants: A Randomized Controlled Trial. Pediatr Crit Care Med. 2017 Sep;18(9):869-875. doi: 10.1097/PCC.0000000000001221. PMID 28617764
- [Background] Fu ZY, Huang C, Lei L, Chen LC, Wei LJ, Zhou J, Tao M, Quan MT, Huang Y. The effect of oropharyngeal colostrum administration on the clinical outcomes of premature infants: A meta-analysis. Int J Nurs Stud. 2023 Aug;144:104527. doi: 10.1016/j.ijnurstu.2023.104527. Epub 2023 May 19. PMID 37295286
- [Background] da Rosa Pereira K, Levy DS, Procianoy RS, Silveira RC. Impact of a pre-feeding oral stimulation program on first feed attempt in preterm infants: Double-blind controlled clinical trial. PLoS One. 2020 Sep 9;15(9):e0237915. doi: 10.1371/journal.pone.0237915. eCollection 2020. PMID 32903261
- [Background] Bashir T, Reddy KV, Kiran S, Murki S, Kulkarni D, Dinesh P. Effect of colostrum given within the 12 hours after birth on feeding outcome, morbidity and mortality in very low birth weight infants: a prospective cohort study. Sudan J Paediatr. 2019;19(1):19-24. doi: 10.24911/SJP.106-1540825552. PMID 31384084